CLINICAL TRIAL: NCT06186115
Title: Intraarticular Gold Microparticles for Hip Osteoarthritis - a 2-year Follow-up Pilot Study.
Brief Title: Intraarticular Gold Microparticles for Hip Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Sten Rasmussen, MD, PhD, Professor Head of Department of Clinical Medicine, Aalborg University, Denmark, Northern Orthopaedic Division, Denmark
Other Study IDs: ArthroGold-6
Record Dates: First submitted 2023-12-16; First posted 2023-12-29 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis, Hip
Keywords: Hip osteoarthritis; Intra articular gold; Outcome
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Gold; Hyaluronic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Gold — Intra articular
  Other Names: Hyaluronic acid

SUMMARY:
In a pilot study, the investigators recently showed that intraarticular metallic gold microparticles reduce knee osteoarthritis pain for up to two years and found associated significant proteomic changes in serum and synovial fluid within eight weeks. This study aim to evaluate the outcome after intra-articular injection of gold microparticles for hip osteoarthritis.

DETAILED DESCRIPTION:
A cohort of 20 patients, aged ≥ 18 years, with pain ≥ 3 months, and Kellgren-Lawrence OA grade 2-4, will beincluded. Metallic gold 20 mg, 72.000 pieces, 20-40 µ-meter (Berlock-Micro-Implants, HumanGoldInject) (1) were injected into the hip joint using hyaluronic acid as the carrier. In total, we treated 24 hip joints. The primary outcome was the Western Ontario and McMaster Universities Arthritis Index (WOMAC).

ELIGIBILITY:
Inclusion Criteria:

* confirmed moderate hip OA (Kellgren-Lawrence grade ≥ 2), pain for more than 3 months, and maximal pain intensity VAS (Visual Analogue Scale, 0-10) ≥ 5 during the last week

Exclusion Criteria:

* exclusion criteria were 1) malignancy, 2) active infection and antibiotic treatment, 3) active treatment with steroids, biological or other anti-rheumatic medication, 4) history of chronic pain condition, 5) inability to comply with the protocol, and 6) inadequacy in written and spoken national language.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Radiographically confirmed moderate hip OA .
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-03-04 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
WOMAC | 2 year
  Western Ontario and McMaster Universities Arthritis Index, sub-scores for pain, stiffness, and function, containing 24 questions: 5 pain questions, two stiffness questions, and 17 physical function questions.

SECONDARY OUTCOMES:
PainDetect | 2 year
  The secondary outcome measure PainDetect questionnaire (PDQ) comprises three major components, gradation of pain, pain course pattern, and radiating pain. Seven questions evaluate the gradation of pain. The patient scored each question using a 0 to 5 score with 0 = never, 1 = hardly noticed, 2 = slightly, 3 = moderately, 4 = strongly and 5 = very strongly. There is one question evaluating pain course patterns. Patients select from one of four pictures indicating which pattern best describes their course of pain. Each picture has a unique score of 0, -1, or +1 (2 pictures have this score possible). One question evaluates radiating pain with a yes (score of +2) or no (score of 0) response option. PDQ is scored from 0 to 38, with total scores < 13 considered to represent nociceptive pain, 13-18 possible neuropathic pain, and > 18 representing neuropathic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Sten Rasmussen, MD PhD, Principal Investigator — Northern ODD
Locations (1):
- Aalborg University Hospital, Aalborg, Region Northern Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Yes
After the publication of the study
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Available after publication
Access Criteria: Will be available at VBN Aalborg University

REFERENCES:
- [Background] Rasmussen S, Kjaer Petersen K, Kristiansen MK, Skallerup J, Aboo C, Thomsen ME, Skjoldemose E, Jorgensen NK, Stensballe A, Arendt-Nielsen L. Gold micro-particles for knee osteoarthritis. Eur J Pain. 2022 Apr;26(4):811-824. doi: 10.1002/ejp.1909. Epub 2022 Feb 1. PMID 35076138
- [Background] Danscher G, Rasmussen S. nanoGold and microGold inhibit autoimmune inflammation: a review. Histochem Cell Biol. 2023 Mar;159(3):225-232. doi: 10.1007/s00418-023-02182-9. Epub 2023 Mar 2. PMID 36864314
- [Background] Rasmussen S, Frederickson C, Danscher G. Inhibition of Local Inflammation by Implanted Gold: A Narrative Review of the History and Use of Gold. J Rheumatol. 2023 May;50(5):704-705. doi: 10.3899/jrheum.221150. Epub 2023 Mar 15. No abstract available. PMID 36921973
- See also: Sten Rasmussen — https://vbn.aau.dk/da/persons/120351